CLINICAL TRIAL: NCT06943118
Title: Comparison of Efficacy of 35% Glycolic Acid vs 20% Salicylic Acid Peel in the Treatment of Post Acne Scars
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hayatabad Medical Complex (Other Government)
Responsible Party: Principal Investigator, Naheed asghar, Associate Professor Dermatology unit HMC, Hayatabad Medical Complex
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hayatabad Medical Complex
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Post Acne Scars
MeSH Terms: interventions — Chemexfoliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 35% glycolic acid peel (Experimental)
  Interventions: Procedure: Chemical Peels
- 20% salicylic acid (Experimental)
  Interventions: Procedure: Chemical Peels

INTERVENTIONS:
Procedure: Chemical Peels — Chemical peel is a dermatological procedure in which chemical solution is applied to the skin to remove the top layer

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two drugs in patients that presents with scars on face after acnes. The effectiveness will be measured by a goodman and baron scale. One group of patients will receive 35% glycolic acid while other group of patients will receive 20% salicylic acid and both groups will be followed by 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-45 years with mild to moderate atrophic post acne scars
* Fitzpatrick skin type 2-4
* No active acne or ongoing systemic acne treatment

Exclusion Criteria:

* Pregnancy and breast feeding
* History of keloid or hypertrophic scars
* Use of retinoids or chemical peel in last 3 months
* Active skin infections
* History of hyperpigmentation after any procedure
* Hypersensitivity to aspirin

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
improvement in acne scars as per Goodman and baron scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: khizar hayat, MBBS, Study Chair — Hayatabad Medical Complex Peshawar, KPK pakistan
Locations (1):
- Hayatabad Medical Complex, Peshawar, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No